CLINICAL TRIAL: NCT07155850
Title: Early Feasibility Clinical Investigation Using a Novel 90-Yttrium-based Internal Radiotherapy Platform, YntraDose™ in Unresectable Locally Advanced Pancreatic Adenocarcinoma (LA-PDAC) as an add-on Therapy to First-line SOC (Chemotherapy)
Brief Title: Early Feasibility Clinical Investigation to Assess YntraDose™ as a Neoadjuvant Treatment for LA-PDAC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: BetaGlue Therapeutics SpA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP-PDAC-25-01
Record Dates: First submitted 2025-08-01; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Pancreatic Ductal Adenocarcinoma (PDAC); Locally Advanced; Unresectable
Keywords: LA-PDAC; Yttrium-90; YntraDose™

STUDY DESIGN:
Intervention Model Description: Multicentre, open-label, prospective, early feasibility clinical investigation to assess the safety, tolerability and feasibility of YntraDose™ treatment following percutaneous administration under US/CT guidance.
Masking Description: No masking for either the patient or user
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- YntraDose™ implantation (Experimental): YntraDose™ is a single use radiotherapy medical device containing Yttrium-90 microspheres administered intratumourally and percutaneously into the pancreas
  Interventions: Device: Medical device containing Y-90 microspheres delivered intratumorally and percutaneously into the pancreas

INTERVENTIONS:
Device: Medical device containing Y-90 microspheres delivered intratumorally and percutaneously into the pancreas — YntraDose™ is a locoregional therapy device used for percutaneous radio-ablation of solid tumours

SUMMARY:
The goal of this clinical investigation is to learn if a new type of radiotherapy works to treat pancreatic cancer that cannot be removed surgically. It will also learn about the safety of the new treatment when combined with chemotherapy. The treatment involves injecting a radioactive implant (medical device) directly into the pancreatic tumour on one occasion only. The main questions it aims to answer are:

* Is the new treatment safe and tolerable when used in combination with standard of care chemotherapy.
* Is it feasible to inject the new treatment directly into a patient's pancreatic tumour.
* What is the impact of this new treatment on a patient's quality of life including a pain evaluation.
* To assess how the pancreatic tumour responds to the treatment during the 3 month follow up.

Participants will:

* Participate in the research study for approximately 7 months and will receive standard of care chemotherapy throughout their participation.
* Participants will initially receive standard of care chemotherapy which will be stopped after 2 months to reassess the tumor by a multidisciplinary tumor board. Chemotherapy will resume and the test device will be administered between chemotherapy treatments. The new treatment involves a single injection of the radioactive implant directly into the pancreatic tumour. Following treatment, the participant's standard of care chemotherapy will resume.
* Participants will attend follow up visits over 3 months.
* Participants will visit the clinic on 8 separate occasions and on one occasions, will remain in hospital for 2 nights/3 days to receive treatment with the new radiotherapy device and to monitor for safety.
* Participants will complete questionnaires to check how the treatment is affecting their daily lives and pain levels.
* Participants will undergo different types of imaging (scans) such as CT, MRI.
* Participants will have bloods and urine taken to monitor safety.

DETAILED DESCRIPTION:
The study is a multicentre, open-label, prospective, early feasibility clinical investigation to assess the safety, tolerability and feasibility of YntraDose™ treatment following percutaneous administration under Ultrasound/CT guidance.

The investigational device is YntraDose™, which is a locoregional therapy device used for percutaneous radio-ablation of solid tumours delivering targeted radiation using Y-90 microspheres injected directly into the tumour site, within a glue matrix holding the Y-90 microspheres in place. The product is designed for single use.

YntraDose™ is indicated as a neoadjuvant therapy and add-on treatment to first-line standard of care therapy in patients with unresectable LA-PDAC. The aim of YntraDose™ development is to combine it with chemotherapy standard of care (FOLFIRINOX or gemcitabine/nab-paclitaxel). Combining systemic chemotherapy with radiotherapy for local disease control, may improve time to progression of local disease, pain control, performance status, and quality of survival, and in a neoadjuvant setting may convert tumours to resectability.

YntraDose™ will be administered intratumorally and percutaneously into the pancreas under ultrasound/CT guidance. The Y-90 microspheres have been designed to deliver a localized distribution of beta radiation within the target tumour. The radiation from these particles causes direct damage to cancer cell DNA, which renders them incapable of further cell division and proliferation, leading to tumour shrinkage. The glue matrix is a hydrogel that polymerizes in the site of implantation and serves to retain the Y 90 radioactive microspheres in-situ facilitating the effect of radioactive microspheres in the tumoural tissue only.

Ten (10) patients with unresectable locally advanced pancreatic ductal adenocarcinoma meeting the eligibility criteria will be recruited into the clinical investigation.

ELIGIBILITY:
Inclusion Criteria (Main):

* Histologically or cytologically proven Pancreatic Adenocarcinoma.
* Stage of disease defined as unresectable Locally Advanced Pancreatic Cancer.
* No prior radiotherapy for pancreatic cancer.
* Target tumour with a minimum diameter of 2.6 cm and a volume of from 9 to 34 ml.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
* Patient has acceptable hematological parameters including white and red blood counts, liver and renal function that makes them suitable to receive SoC chemotherapy as per local clinical practice.
* Life expectancy of ≥6 months at screening.

Exclusion Criteria (Main):

* Evidence of distant metastases based on the restaging process after two months of induction chemotherapy identified using CT/MRI/18 FDG PET assessment.
* Evidence of switch from unresectable status to resectable status of disease after two months of induction chemotherapy.
* More than one primary lesion, if one of the primary lesions is not a good candidate for debulking with YntraDose™, due to clinical reasons and/or decision made by the local MDTB.
* ECOG is higher than 1.
* History of malignancy in the last 3 years.
* Blood clotting disorders (INR > 1.5, PLT < 50,000/µl - risk of bleeding during organ puncture).
* Active systemic or local infection (e.g. peritonitis, abscess).
* Severe organ failure (e.g. end-stage liver, kidney, heart failure).
* Cardiological and other diseases that threaten the use of anesthesia.
* Pancreatitis (acute or exacerbation of chronic inflammation).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability assessment | From commencement of induction chemotherapy (immediately following screening) to the end of the follow up period at 3 months.
  The primary endpoint is safety and tolerability and will be measured by the frequency of treatment-emergent adverse events (TEAEs), graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE, v5.0).
Feasibility of administration of the medical device | From implantation of the medical device to the end of the follow up period at 3 months.
  To evaluate the feasibility of YntraDose™ percutaneous administration under US/CT guidance for implant in the target tumour lesion, without major clinical complications defined as needing medical intervention to resolve any significant adverse event or medical issue arising from the administration of YntraDose™.

SECONDARY OUTCOMES:
Patient Quality of Life | From enrollment to the end of the follow up period at 3 months.
  To evaluate the patient's quality of life using the EORTC QLQPAN26 assessment questionnaire, for people with pancreatic ductal adenocarcinoma (PDAC).
Pain Assessment | Pain assessments will be collected during the 2 pre-implantation screening visits and at 1 week, 1 month, 2 months and 3 months following implantation of the investigational device.
  Pain will be assessed using a 11-point NPRS (Numerical Pain Rating Scale). collected at screening and during the follow up period.
Patient tumour response following treatment with the medical device | From baseline assessments to the end of the follow up period at 3 months.
  To evaluate the change in the tumour marker carbohydrate antigen (CA) 19-9 levels comparing baseline levels to the (CA) 19-9 levels at follow up.
Metabolic tumour response evaluation | From baseline to the to the end of the follow up period at 3 months.
  Metabolic tumour response according to [18F]2-fluoro-2-deoxy-Dglucose positron emission tomography (18F-FDG-PET) will be measured at baseline and subsequent follow-up time points, for total lesion glycolysis (TLG), standardised uptake values SUVMax and SULMax, target tumour volume change as imaged by CT scans.

IPD SHARING:
Plan to Share IPD: Yes
A Clinical Investigation Report will be prepared according to ISO 14155:2020 (Annex D) and UNI EN ISO 14155:2025. The report will be a record of the investigation conduct and findings and will be subject to approval by the Investigators who will sign the final report. Patient data will be analyzed collectively in accordance with the investigation Statistical Analysis Plan. Individual patients will not be identified in any report, presentation or publication resulting from the study.
Supporting Information: CSR
Time Frame: As required, a copy of the final Clinical Investigation Report and a summary of the results written in a manner that is understandable to lay persons, will be provided to the Regulatory Authority and/or Ethics Committee responsible for each participating site within 1 year (12 months) from study completion.
Access Criteria: Regulatory Authorities and/or Ethics Committees responsible for each investigational site will receive the clinical investigation report and lay person summary.
  Results will be posted on clinicaltrials.gov which is a publicly accessible database, 12 months following study completion.